CLINICAL TRIAL: NCT03932110
Title: The Prevalence of Metabolic Syndrome in Patients With Psoriasis and Psoriatic Arthritis and Its Correlation With Disease Severity and Serum Omentin-1 and Visfatin Levels
Brief Title: Metabolic Syndrome in Psoriasis and Psoriatic Arthritis and Correlation With Serum Omentin and Visfatin Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Deniz Dağdelen, M. D., Istanbul Medeniyet University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DDagdelen
Record Dates: First submitted 2019-04-24; First posted 2019-04-30 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Psoriasis Vulgaris; Psoriatic Arthritis; Metabolic Syndrome
Keywords: psoriasis vulgaris; psoriatic arthritis; metabolic syndrome; omentin; visfatin
MeSH Terms: conditions — Arthritis, Psoriatic; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- psoriasis vulgaris, (Other): patients who have only psoriasis vulgaris
  Interventions: Diagnostic Test: omentin, visfatin
- psoriatic arthritis (Other): patients who have psoriatic arthritis
  Interventions: Diagnostic Test: omentin, visfatin
- healthy control (Other): healthy people
  Interventions: Diagnostic Test: omentin, visfatin

INTERVENTIONS:
Diagnostic Test: omentin, visfatin — diagnostic blood test

SUMMARY:
In this study, the prevalence of metabolic syndrome in psoriatic and psoriatic arthritis patients as well as the parameters of metabolic syndrome will be examined. At the same time, the levels of omentin and visfatin adipokines associated with metabolic syndrome and obesity will be measured by measuring the disease severity (by PASI psoriasis, clinical activity score for psoriatic arthritis). The patients who accepted to participate in the study , who were admitted to the dermatology outpatient clinic were included in the study. For the blood tests required after the examination, 2 tubes of blood will be taken for the measurement of omentin and visfatin. 80 psoriasis, 40 psoriatic arthritis and 60 healthy volunteers were planned to be studied. AHA / NHLBI, 2005 (revised ATP III criteria) criterion for the diagnosis of metabolic syndrome will be used. Omentin and visfatin levels are compared with the severity of the disease for psoriasis and psoriatic arthritis, and it will be examined whether it is proinflammatory or antiinflammatory.

ELIGIBILITY:
Inclusion Criteria:

1. Patients followed up for psoriasis and psoriatic arthritis in dermatology and rheumatology clinic
2. Patients older than 18 years
3. Patients who accept dermatological and rheumatic examination
4. Patients not receiving systemic treatment related to the disease in the last 1 month

Exclusion Criteria:

1. Patients with autoimmune and rheumatic diseases other than psoriasis and psoriatic arthritis
2. Patients under 18 years
3. Patients who do not accept dermatological and rheumatic examination Patients receiving systemic therapy for the last 1 month pregnant and nursing moms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
omentin | 6 months
  Omentin (omentin 1-2) is a specific protein that consists of amino acids released from vascular vessels
visfatin | 6 months
  Visfatin is an insulin-like protein that binds to insulin receptors produced mostly from visceral fatty tissue.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medeniyet University, Department of dermatology, Istanbul
  - Istanbul Medeniyet University, Istanbul

IPD SHARING:
Plan to Share IPD: No